CLINICAL TRIAL: NCT00550966
Title: Efficacy of a Psychoeducative Program for Improving Quality of Life in Fibromyalgic Patients [Study Protocol]
Acronym: FIBRO-Qol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institut Catala de Salut (Other Government)
Collaborators: Agència d'Avaluació de Tecnologia i Recerca Mèdiques (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 077/25/2006
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Quality of life; Primary Care; Non-pharmacological treatment; Cost / Cost-efficacy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Randomized controlled trial with a 12-month follow-up involving two groups, one of which is the intervention group that includes patients receiving a psychoeducative program and the other is the control group formed by patients treated for FM in the usual way.
  Setting. Three urban PC centers in the province of Barcelona (Spain) Sample. The total sample comprises 218 patients (over 18 years of age) suffering FM, selected from a database (Rheumatology service-Viladecans hospital) of patients with this illness. Only those patients introduced in the database between the years 2005 and 2007 are included in the selection. Selected patients are asked for written informed consent to participate in the study.
  Interventions: Behavioral: Psychoeducative program in fibromyalgic patients

INTERVENTIONS:
Behavioral: Psychoeducative program in fibromyalgic patients — Multi-component program including information about the illness, counselling about physical exercise and training in autogenic relaxation. The intervention consists on nine 2 hour sessions delivered during a two month period. The pharmacological treatment prescribed by the physician is maintained in both groups.
  Other Names: Fibromyalgia; Psychoeducative program

SUMMARY:
This research project pretends to demonstrate that a psychoeducative program implemented in the context of PC can produce a significant increase in the quality of life of patients with FM, as well as a decrease in the use of sanitary and social services, compared to usual care.

DETAILED DESCRIPTION:
Most fibromyalgic patients are attended at primary care (PC). However, the effectiveness of the treatments prescribed by general practitioners is usually scarce. The main objective of the present research is to assess the efficacy of a structured psychoeducative intervention, combined with relaxation, developed to improve the quality of life of patients suffering fibromyalgia (FM). The second objective is to assess the cost-effectiveness of this multimodal intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aged between 18-75 years-old who meet the diagnostic criteria of fibromyalgia established by the American College of Rheumatology (ACR)

Exclusion Criteria:

* Patients with a diagnosis not based on the ACR criteria
* Those with cognitive impairment or suffering from physical mental/psychiatric limitations
* Severe concurrent rheumatologic illness that impede participation in the study evaluations
* Those who are not expected to live at least 12 months
* Those without schooling.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2007-09; Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life is measured with the FIQ and the EuroQol-5D. | 1, 2, 6 and 12 months later

SECONDARY OUTCOMES:
The use of sanitary services is measured with an adapted version of the Client Service Receipt Inventory (CSRI) | 1, 2, 6 and 12 months later

CONTACTS AND LOCATIONS:
Overall Officials: Rita Fernández-Vergel, Doctor, Principal Investigator — Institut Català de Salut (ICS); María Teresa Peñarrubia, Doctor, Study Director — Institut Català de Salut (ICS); Elena Blanco, Doctor, Study Chair — ICS; Mónica Jiménez, Doctor, Study Chair — ICS; Adrián Montesano, psychology, Study Director — Fundació Jordi Gol i Gurina. ICS; Antonio Serrano, psychiatrist, Study Director — Sant Joan de Déu-Serveis de Salut Mental; Juan Vicente Luciano, psychology, Study Chair — Red de Investigación en Actividades Preventivas y Promoción de la Salud en Atención Primaria (RedIAPP); Mª del Camino Verduras, Doctor, Study Chair — ICS; José Miguel Ruíz, Reumatology, Study Chair — ICS
Locations (1):
- ABS Bartomeu Fabres Anglada. Institut Català de Salut., Gavà, Barcelona, Spain

REFERENCES:
- [Derived] Luciano JV, Sabes-Figuera R, Cardenosa E, T Penarrubia-Maria M, Fernandez-Vergel R, Garcia-Campayo J, Knapp M, Serrano-Blanco A. Cost-utility of a psychoeducational intervention in fibromyalgia patients compared with usual care: an economic evaluation alongside a 12-month randomized controlled trial. Clin J Pain. 2013 Aug;29(8):702-11. doi: 10.1097/AJP.0b013e318270f99a. PMID 23328339
- [Derived] Luciano JV, Martinez N, Penarrubia-Maria MT, Fernandez-Vergel R, Garcia-Campayo J, Verduras C, Blanco ME, Jimenez M, Ruiz JM, Lopez del Hoyo Y, Serrano-Blanco A; FibroQoL Study Group. Effectiveness of a psychoeducational treatment program implemented in general practice for fibromyalgia patients: a randomized controlled trial. Clin J Pain. 2011 Jun;27(5):383-91. doi: 10.1097/AJP.0b013e31820b131c. PMID 21317775